CLINICAL TRIAL: NCT03318185
Title: Efficacy and Safety of Gasless Single-port Laparoscopic-assisted Radical Resection for Rectal Carcinoma
Brief Title: Gasless Single-port Laparoscopic-assisted Radical Resection for Rectal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017140
Record Dates: First submitted 2017-09-20; First posted 2017-10-23 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Laparoscopic Surgery
Keywords: gasless single-port laparoscopic surgery;rectal carcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gasless single-port laparoscopic surgery (Experimental): radical resection of rectal carcinoma is performed by gasless single-port laparoscopic-assisted surgery.
  Interventions: Procedure: gasless single-port laparoscopic surgery
- conventional laparoscopic surgery (Sham Comparator): radical resection of rectal carcinoma is performed by conventional laparoscopic surgery.
  Interventions: Procedure: conventional laparoscopic surgery

INTERVENTIONS:
Procedure: gasless single-port laparoscopic surgery — The single-port laparoscopic surgery is performed when the maneuvering room is provided by external suspension system.
  Arms: gasless single-port laparoscopic surgery
Procedure: conventional laparoscopic surgery — The multi-port laparoscopic surgery is performed when the belly is inflated with carbon dioxide to provide maneuvering room.
  Arms: conventional laparoscopic surgery

SUMMARY:
This project aims to investigate the safety and effectiveness of gasless single-port laparoscopic-assisted radical resection (GSLR) in the treatment of rectal carcinoma.

DETAILED DESCRIPTION:
The gasless single-port laparoscopic-assisted surgery (GSLS) is associated with rapid recovery and shorter postoperative hospital stay and no pneumoperitoneum complications occur after the operation. To our knowledge, there have been no reports about GSLS applied to the treatment of gastrointestinal cancer in the world. To explore the safety and effectiveness of GSLS in rectal cancer patients, this project plans to evaluate the operation time, cardio-pulmonary function, postoperative pain, immunologic function and restoration of bowel function after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Rectal carcinoma;The distance between tumor and anal verge is 5-15cm; The primary tumor can radical resect.

Exclusion Criteria:

* Neoadjuvant therapy;Surgical contraindication.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function | Change from baseline PaO2/FiO2 ratio 10 minutes after the surgery is over.
  Estimate the pulmonary function in the perioperational period by blood gas analysis, which will be compared with comparator.The main parameter partial pressure of oxygen(PaO2)/inspired oxygen fraction(FiO2) ratio is the ratio of arterial oxygen partial pressure to fractional inspired oxygen.
Immunologic function | Change from baseline CD4/CD8 ratio 7 days after operation.
  Estimate the immunologic function in the perioperational period by blood lymphocyte analysis, which will be compared with comparator.The main parameter cluster of differentiation 4(CD4)/cluster of differentiation 8(CD8) ratio is the ratio of lymphocyte CD4 numbers to lymphocyte CD8 numbers.

SECONDARY OUTCOMES:
Operation time | at 1 day
  Measure the operation time, which will be compared with comparator.
Postoperative pain | 72 hours after operation
  Measure the postoperative pain after operation by numerical rating scale(NRS), which will be compared with comparator.
Bowel function | up to 1 week after operation
  Measure the restoration of bowel function after operation, which will be compared with comparator.The bowel function was evaluated by first flatus.
Number of the lymph node dissection | at 1 week after operation
  Measure the number of the regional lymph node dissection after operation, which will be compared with comparator.

CONTACTS AND LOCATIONS:
Overall Officials: Jijian Wang, phD, Study Chair — The Second Affiliated Hospital of Chongqing Medical University; Yaxu Wang, phD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Yang Li, phD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Daihua Zhu, phD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Jianbo Zhang, phD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Haitao Gu, phD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Shiji Zhou, phD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Zhiquan Xu, Bachelor, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- Gastrointestinal Surgery Department of the Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No